CLINICAL TRIAL: NCT00635518
Title: Randomized Controlled Trial of Dietary Advice in Primary Care to Promote Healthy Feeding of Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was canceled and no resources are available.
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Marcia Regina Vitolo, PhD, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: vitolo1
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Breast Feeding
Keywords: Health Plan Implementation; Feeding and Eating Disorders of Childhood; Breast Feeding; Overweight; Child; Infant Nutrition Physiology; Public Health
MeSH Terms: conditions — Breast Feeding; Feeding and Eating Disorders of Childhood; Overweight

STUDY DESIGN:
Intervention Model Description: Study Withdrawn
Oversight: Data Monitoring Committee: No

ARMS (1):
- I, Intervention (Other)
  Interventions: Behavioral: Ten Steps for Healthy Feeding children programme

INTERVENTIONS:
Behavioral: Ten Steps for Healthy Feeding children programme — Ten Steps for Healthy Feeding children
  Other Names: Infant Nutrition Programme

SUMMARY:
A cluster randomized field trial to evaluate the impact that training healthcare workers in healthy feeding practices has on the nutrition and health of children.

DETAILED DESCRIPTION:
A cluster randomized controlled trial. Twenty health care service sites were randomly assigned to the intervention or control groups. Health care workers of the intervention health care service sites received training based on the programme "Ten steps for healthy feeding for children from birth to two years old".

Pregnant women, in their third term, were enrolled in the study. At 6 and 12 months of age, the mothers were interviewed at home using a semi-structured questionnaire with pre-coded close- and open-ended questions and the children were evaluated.

ELIGIBILITY:
Inclusion Criteria:

- All pregnant women in the last quarter of the gestation.

Exclusion Criteria:

* HIV-positive mothers
* congenital malformation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Márcia R Vitolo, postdoctoral, Principal Investigator — Federal University of Health Sciences of Porto Alegre